CLINICAL TRIAL: NCT03500445
Title: Open-label, Single-arm, Phase 2 Study of Initial Treatment With Daratumumab (Darzalex), Carfilzomib (Kyprolis), Lenalidomide (Revlimid) and Low Dose Dexamethasone (DKRd) in Newly Diagnosed, Multiple Myeloma Requiring Systemic Chemotherapy
Brief Title: Daratumumab, Carfilzomib, Lenalidomide and Low Dose Dexamethasone (DKRd) in Newly Diagnosed, Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-1097
Record Dates: First submitted 2018-04-09; First posted 2018-04-18 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Myeloma; Multiple Myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell; Multiple Myeloma | interventions — daratumumab; carfilzomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (D-KRd) (Experimental)
  Interventions: Drug: Daratumumab; Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab — Daratumumab (16 mg/kg) will be administered as an IV infusion:
  * Cycle 1-2: 16 mg/kg weekly
  * Cycles 3-8: 16 mg/kg IV infusion every 2 weeks
  * Cycles 9-24: 16 mg/kg IV infusion Day 1
  Other Names: DARZALEX®
Drug: Carfilzomib — Carfilzomib will be given as an IV infusion over 30 minutes:
  * Cycle 1: 20 mg/m2 Days 1, 2; 36 mg/m2 Days 8, 9, 15, 16. Alternatively, intermediate dose escalation (to 27mg/m2 on days 8, 9 of cycle 1) will be allowed at the treating physician's discretion.
  * Cycle 2-9: 36 mg/m2 (or best tolerated dose) Days 1, 2, 8, 9, 15 and 16
  * Cycles 9-24: 36 mg/m2 (or best tolerated dose) Days 1, 2, 15 and 16
  Other Names: KYPROLIS®
Drug: Lenalidomide — Lenalidomide will be taken orally as follows:
  • Cycles 1-24: 25 mg (or best tolerated dose) PO Days 1-21
  Other Names: REVLIMID®
Drug: Dexamethasone — Dexamethasone will be administered prior to carfilzomib (on days that they coincide), as follows:
  * Cycles 1-9: 40 mg PO (subjects ≤ 75 years) or 20 mg PO (subjects ≥ 75 years) per week
  * Cycles 9-24: 20 mg PO per week
  During weeks when daratumumab is given: 40 mg dexamethasone weekly, 20 mg prior to daratumumab infusion and 20 mg PO the day after
  During weeks with no daratumumab, single dose of 20 mg on day 1

SUMMARY:
The purpose of this study is to determine response rate after 8 cycles of D-KRd (daratumumab, carfilzomib, lenalidomide (Revlimid) and dexamethasone in patients with multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, previously untreated myeloma requiring systemic chemotherapy

  • Prior treatment of hypercalcemia or spinal cord compression or active and/or aggressively progressing myeloma with corticosteroids or lenalidomide or bortezomib-based regimens does not disqualify the patient (the treatment dose should not exceed the equivalent of 160 mg of dexamethasone in a 4 week period or not more than 1 cycle of Proteasome Inhibitor / Immunomodulatory-based therapy)
* Both transplant and non-transplant candidates are eligible.
* Diagnosis of symptomatic multiple myeloma as per current International Myeloma Working Group (IMWG) uniform criteria prior to initial treatment
* Monoclonal plasma cells in the Bone Marrow (BM) ≥ 10% or presence of a biopsy-proven plasmacytoma
* Measurable disease, prior to initial treatment as indicated by one or more of the following:

  * Serum M-protein ≥ 1 g/dL
  * Urine M-protein ≥ 200 mg/24 hours
  * If serum protein electrophoresis is felt to be unreliable for routine M-protein measurement, then quantitative immunoglobulin levels are acceptable
  * Serum freelite measurable disease as per current IMWG criteria
* Bone marrow specimen will be required at study entry; available DNA sample from pre-induction BM will be used for calibration step for MRD evaluation by gene sequencing.
* Males and females ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Adequate hepatic function, with bilirubin ≤ 1.5 x upper limit of normal (ULN) and aspirate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x ULN
* Absolute Neutrophil Count (ANC) ≥ 1.0 x 109/L, hemoglobin ≥ 8 g/dL, platelet count ≥ 75 x 109/L.
* Calculated creatinine clearance (by Cockroft-Gault) ≥ 50 mL/min or serum creatinine below 2 g/dL
* Woman of childbearing potential must have 2 negative pregnancy tests prior to initiating lenalidomide.
* Woman of childbearing potential must agree to use 2 reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) for at least 28 days before starting lenalidomide; 2) while participating in the study; and 3) for at least 30 days after discontinuation from the study.
* Male subjects must agree to use a latex condom during sexual contact with females of childbearing potential while participating in the study and for at least 90 days following discontinuation from the study even if he has undergone a successful vasectomy.
* All study participants in the US must be consented to and registered into the mandatory Revlimid Risk Evaluation and Mitigation Strategy (REMS®) program and be willing and able to comply with the requirements of Revlimid REMS®.
* Voluntary written informed consent.

Exclusion Criteria:

* Frail non-transplant candidates, defined as in Palumbo et al, Blood 2015.
* Non-secretory or hyposecretory multiple myeloma, prior to initial treatment defined as <1.0 g/dL M-protein in serum, <200 mg/24 hr urine M-protein, and no measurable disease as per IMWG by Freelite.
* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Amyloidosis
* Plasma cell leukemia
* Waldenström's macroglobulinemia or Immunoglobulin M-producing (IgM) myeloma
* Radiotherapy to multiple sites or immunotherapy within 4 weeks before start of protocol treatment (localized radiotherapy to a single site at least 1 week before start is permissible)
* Participation in an investigational therapeutic study within 3 weeks or within 5 drug half-lives (t1/2) prior to first dose, whichever time is greater
* Potential subjects with evidence of progressive disease as per IMWG criteria
* Patients not able to tolerate daratumumab, carfilzomib, lenalidomide or dexamethasone
* Peripheral neuropathy ≥ Grade 2 at screening
* Diarrhea > Grade 1 in the absence of antidiarrheals
* Central Nervous System (CNS) involvement
* Pregnant or lactating females
* Major surgery within 3 weeks prior to first dose.
* Myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Prior or concurrent pulmonary embolism
* Known moderate or severe persistent asthma or known chronic obstructive pulmonary disease (COPD)

  * Known or suspected chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal
  * Moderate or severe persistent asthma within the past 2 years, or currently has uncontrolled asthma of any classification. Note that subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed in the study.
* Rate-corrected QT interval of electrocardiograph (QTc) > 470 msec on a 12-lead ECG during screening
* Uncontrolled hypertension or diabetes
* Acute infection requiring systemic antibiotics, antivirals, or antifungals within two weeks prior to first dose
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.
* Non-hematologic malignancy or non-myeloma hematologic malignancy within the past 3 years except a) adequately treated basal cell, squamous cell skin cancer, thyroid cancer, carcinoma in situ of the cervix, or prostate cancer < Gleason Grade 6 with stable prostate specific antigen levels or cancer considered cured by surgical resection alone
* Any clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-02-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of stringent complete response (sCR) | 8 months
Rate of minimal residual disease (MRD)-negative disease as assessed by Next Generation Sequencing | 8 months

SECONDARY OUTCOMES:
Long term rate of MRD-negative disease | 2 years
Duration of response | 1 year
Rate of progression free survival | 2 years
Time to progression | 2 years
Overall survival rate | 2 years
Overall response rate | 2 years
Number of grade 2 or higher side effects as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 criteria | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Jakubowiak, MD, PhD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided